CLINICAL TRIAL: NCT04663087
Title: A Pilot Randomized Clinical Trial of the XSTAT Hemostatic Device in the Prehospital Setting
Brief Title: Feasibility of Evaluating XSTAT Use in the Prehospital Setting
Acronym: PhoXSTAT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor stopped enrollment
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Jan O. Jansen, Primary Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-300003647
Record Dates: First submitted 2019-10-07; First posted 2020-12-10 (Actual); Results first posted 2024-12-11 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-12

CONDITIONS: Shock, Hemorrhagic; Injury Penetrating; Hemorrhage
Keywords: hemorrhagic shock; hemostatic sponge; penetrating injury; junctional wounds; prehospital
MeSH Terms: conditions — Shock, Hemorrhagic; Wounds, Penetrating; Hemorrhage | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Treatment with XSTAT (Experimental): Participants randomized to the treatment arm will be treated using the study device - XSTAT.
  Interventions: Device: XSTAT
- Standard Care (Other): Participants assigned to the control group receive standard prehospital care, consisting of direct pressure/dressings.
  Interventions: Other: Standard of Care

INTERVENTIONS:
Device: XSTAT — XSTAT application will follow the manufacturer's guidance, with injection into bleeding junctional wounds. A sufficient number of sponges are used to fill the injury void. Repeated XSTAT application is performed in the event of persistent bleeding. The trial packs will contain two devices.
  Other Names: XSTAT 12
  Arms: Treatment with XSTAT
Other: Standard of Care — As currently provided by EMS services
  Arms: Standard Care

SUMMARY:
This study evaluates the prehospital use of the XSTAT device to control bleeding in junctional wounds. Participants will be randomized to the use of XSTAT versus standard care.

DETAILED DESCRIPTION:
The XSTAT® device injects small, rapidly-expanding cellulose sponges into the wound cavity using a syringe-like delivery system. In the wound, XSTAT® sponges expand and swell to fill the wound cavity, within 20 seconds of contact with blood, facilitating compression of bleeding structures. XSTAT® can be applied through skin wounds. The system can readily access deep vascular structures. While rapidly hemostatic, the hemostatic sponges are also relatively easy to remove. In the setting of junctional bleeding, XSTAT® may allow for hemostatic pressure generation from within the wound tract rather than from external compression (as with a tourniquet or manual compression).

Hemorrhage should be controlled as early as possible, ideally before reaching a trauma center or medical treatment facility. Given its small size, low weight, and ease of application, the XSTAT® device is well-suited for prehospital use, in both the civilian and military setting, and this is probably where the device's applicability lies.

The investigators anticipate that a full-scale trial will be conducted based on the questions this pilot study addresses, including the following:

1. the number of penetrating junctional zone injuries encountered in the prehospital civilian setting.
2. the feasibility of randomizing patients in the prehospital setting.
3. usability.
4. safety.
5. validation of the proposed primary outcome of an efficacy trial.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥15 years or estimated body weight ≥50 kg.
2. Penetrating junctional injury (femoral or axillary), with i. visible bleeding ii. too proximal to be controlled with a tourniquet
3. Patient will be taken to participating level I trauma center, directly from the scene

Exclusion Criteria:

1. Prisoners, children <15 years old, known pregnant patients.
2. Patients receiving chest compressions (prior to XSTAT® use).
3. Patients with an opt-out bracelet.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2022-10-29 (Actual); Primary Completion 2023-06-21 (Actual); Study Completion 2023-08-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jan Jansen, MBBS, PhD, Principal Investigator — The University of Alabama at Birmingham
Locations (1):
- UAB Hospital, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Stephens SW, Farley P, Collins SP, Wong MD, Panas AB, Dennis BM, Richmond N, Inaba K, Brown KN, Holcomb JB, Jansen JO. Multicenter social media community consultation for an exception from informed consent trial of the XStat device (PhoXStat trial). J Trauma Acute Care Surg. 2022 Feb 1;92(2):442-446. doi: 10.1097/TA.0000000000003425. PMID 34620774

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a pilot/feasibility trial. The trial was conducted in the prehospital setting, and was an Exception From Informed Consent (EFIC) study. Patients were to be enrolled by EMS agencies. Only one patient was enrolled.
Period: Overall Study
Arm/Group | Treatment With XSTAT | Standard Care
Started | 0 | 1
Completed | 0 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Only one patient was enrolled; additional data not provided to preserve confidentiality
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment With XSTAT | Standard Care | Total
Number analyzed (Participants) | 0 | 1 | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years |  | 0 | 0
  Between 18 and 65 years |  | 1 | 1
  >=65 years |  | 0 | 0
Sex/Gender, Customized [Count of Participants; unit: Participants] |  | NA — Data not provided to preserve confidentiality | NA — Total not calculated because data are not available (NA) in one or more arms.
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Patients With Hemorrhage From Junctional Wounds
Description: The investigators will track the number of junctional wounds that are treated by participating EMS personnel versus the number of participants who were enrolled in this study. This will help the investigators understand how many wounds of this type happen, and how many would possibly benefit from the use of the XSTAT device.
Time Frame: Each participant was assessed at the time of arrival in hospital
Population: Only 1 patient enrolled
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment With XSTAT | Standard Care
Number analyzed (Participants) | 0 | 1
Participants | 0 | 1

2. Primary Outcome: Record Blood Lactate Level Result
Description: Record results of routine test
Time Frame: Baseline - on admission
Population: Only 1 patient enrolled
Measure: Number; unit: mmol/l
Arm/Group | Treatment With XSTAT | Standard Care
Number analyzed (Participants) | 0 | 1
mmol/l |  | 3.5

3. Primary Outcome: Base Deficit (mmol/l)
Description: Base excess and base deficit refer to an excess or deficit, respectively, in the amount of base present in the blood. The value is usually reported as a concentration in units of mEq/L (mmol/L), with positive numbers indicating an excess of base and negative a deficit. A typical reference range for base excess is -2 to +2 mEq/L. It is a test performed on a blood sample, venous or arterial. In trauma patients, a metabolic acidosis is indicative of the degree of shock, causing hypoperfusion. A more negative value indicates more severe acidosis, and more severe shock.
Time Frame: Baseline - on admission
Population: Only 1 patient enrolled
Measure: Number; unit: mmol/l
Arm/Group | Treatment With XSTAT | Standard Care
Number analyzed (Participants) | 0 | 1
mmol/l |  | -2.1

4. Primary Outcome: Record Hemoglobin/Hematocrit Result
Description: Record results of routine test
Time Frame: Baseline - on admission
Population: Only 1 patient enrolled
Measure: Number; unit: g/dL
Arm/Group | Treatment With XSTAT | Standard Care
Number analyzed (Participants) | 0 | 1
g/dL |  | 12.7

5. Primary Outcome: Record Platelet Count Result
Description: Record results of routine test
Time Frame: Baseline - on admission
Population: Only 1 patient enrolled
Measure: Number; unit: 10^9 platelets/L
Arm/Group | Treatment With XSTAT | Standard Care
Number analyzed (Participants) | 0 | 1
10^9 platelets/L |  | 267

6. Primary Outcome: Record Prothrombin Time Result
Description: Record results of routine test
Time Frame: Baseline - on admission
Population: Only 1 patient enrolled
Measure: Number; unit: seconds
Arm/Group | Treatment With XSTAT | Standard Care
Number analyzed (Participants) | 0 | 1
seconds |  | 13.8

7. Primary Outcome: Record International Normalized Ratio (INR) Result
Description: Record results of routine test
Time Frame: Baseline - on admission
Population: Only 1 patient enrolled
Measure: Number; unit: Ratio
Arm/Group | Treatment With XSTAT | Standard Care
Number analyzed (Participants) | 0 | 1
Ratio |  | 1.1

8. Primary Outcome: Record Activated Partial Thromboplastin Time (APTT) / Ratio Result
Description: Record results of routine test
Time Frame: Baseline - on admission
Population: Only 1 patient enrolled
Measure: Number; unit: seconds
Arm/Group | Treatment With XSTAT | Standard Care
Number analyzed (Participants) | 0 | 1
seconds |  | 27

9. Primary Outcome: Record Thromboelastograph (TEG) Result if Available
Description: Record results of routine test
Time Frame: Baseline - on admission
Population: Only 1 patient enrolled, who did not have this test done (which was not mandatory).
Arm/Group | Treatment With XSTAT | Standard Care
Number analyzed (Participants) | 0 | 0

10. Primary Outcome: Record Thromboelastogram (ROTEM) Result if Available
Description: Record results of routine test
Time Frame: Baseline - on admission
Population: Only 1 patient enrolled, who did not have this test done (which was not mandatory).
Arm/Group | Treatment With XSTAT | Standard Care
Number analyzed (Participants) | 0 | 0

11. Primary Outcome: Ease of Use of XSTAT Device by EMS Personnel
Description: To answer the question "Is the XSTAT device easy to use in the prehospital setting," the study case report forms capture whether EMS personnel found the device easy to insert into a wound, whether the sponges were expelled from the device easily, and whether the EMS personnel were satisfied or dissatisfied with the XSTAT device itself.
Time Frame: From baseline to 29 months (enrollment phase)
Population: Only 1 patient enrolled, randomized to control arm
Arm/Group | Treatment With XSTAT | Standard Care
Number analyzed (Participants) | 0 | 0

12. Primary Outcome: Sponge Removal: Surgeon Opinion of Ease of Removal, Time Required to Remove Sponges, Use of X-rays, Whether Surgeon Was Satisfied or Dissatisfied With the XSTAT Device.
Description: Case report forms capture whether sponges were easy to remove, how much time was required to remove the sponges, whether x-rays were obtained to ensure that no sponges were left in the body, and whether the surgeon was satisfied or dissatisfied with the XSTAT device
Time Frame: From baseline to 29 months (enrollment phase)
Population: Only 1 patient enrolled, randomized to control arm
Arm/Group | Treatment With XSTAT | Standard Care
Number analyzed (Participants) | 0 | 0

13. Primary Outcome: Adverse Events From Use of XSTAT Device
Description: All AEs, whether expected or unexpected will be recorded and reviewed throughout the trial. Each AE will be reported separately, with a description of the event, whether it was related to the device, whether it was serious, and whether it was expected or unexpected.
Time Frame: Randomization through first 7 days, unless discharged earlier
Population: Only 1 patient enrolled, randomized to control arm
Arm/Group | Treatment With XSTAT | Standard Care
Number analyzed (Participants) | 0 | 0

14. Primary Outcome: Survival at 30 Days
Description: Time of death, or survival at 30 days will be recorded
Time Frame: Hospital admission through 30 days
Population: Only 1 patient enrolled
Measure: Number; unit: participants
Arm/Group | Treatment With XSTAT | Standard Care
Number analyzed (Participants) | 0 | 1
participants |  | 1

ADVERSE EVENTS:
Time Frame: From admission to the level 1 trauma center until time of discharge from the level 1 trauma center, typically 28 days.
Description: Standard definitions
Arm/Group | Treatment With XSTAT | Standard Care
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/1
Other Adverse Events (participants affected / at risk) | 0/0 | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2021-05-23): https://cdn.clinicaltrials.gov/large-docs/87/NCT04663087/Prot_001.pdf